CLINICAL TRIAL: NCT05151926
Title: Limb Injuries and Post Injury Rehabilitation Trials - Tibial Shaft Fracture (LIMPER-TSF): a Protocol for Prospective, Randomized,Multicentre Trial Comparing the Early Partial and Early Full Weightbearing After Nailed Tibial Shaft Fracture
Brief Title: Limb Injuries and Post Injury Rehabilitation Trials - Tibial Shaft Fracture
Acronym: LIMPER-TSF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Aleksi Reito, Associate professor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21010
Record Dates: First submitted 2021-10-22; First posted 2021-12-09 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Tibia Fracture
Keywords: intramedullary nail; weight-bearing
MeSH Terms: conditions — Tibial Fractures | interventions — Partial Weight-Bearing; Fracture Fixation, Intramedullary

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full weight-bearing (Experimental): Full immediate weight-bearing postoperatively
  Interventions: Procedure: Full weight-bearing; Procedure: Intramedullary nailing
- Partial-weight bearing (Active Comparator): Partial weight-bearing for the first 6 weeks postoperatively.
  Interventions: Procedure: Partial weight-bearing; Procedure: Intramedullary nailing

INTERVENTIONS:
Procedure: Full weight-bearing — Instruction for full and immediate weight-bearing postoperatively
  Arms: Full weight-bearing
Procedure: Partial weight-bearing — Instruction for partial weight-bearing for 6 weeks postoperatively
  Arms: Partial-weight bearing
Procedure: Intramedullary nailing — Intramedullary nailing of the fractured tibial shaft.

SUMMARY:
Aim of our study is to compare immediate full weight-bearing and partial weight-bearing for 6 weeks after a tibial shaft fracture treated with intramedullary nailing. Co-primary outcome is return to work and physical component scale in the SF-36 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* AO/OTA 42-A/B acute, noncomminuted diaphyseal fracture of the tibia treated with intramedullary nailing with or without posterior malleolus screw fixation
* operated within 72 hours of admittance
* age between 18-65 years

Exclusion Criteria:

* the inability to fill out the Finnish versions of the questionnaires
* previous arthroplasty of the knee or the ankle of the fractured limb
* previous ipsilateral below-knee fracture requiring surgical treatment or ankle arthrodesis
* inability to co-operate
* not living independently (institutionalized living before fracture)
* open fracture (Gustilo grade 2 or over)
* pathologic or stress fracture
* multiple fractures requiring operative treatment in polytrauma patient
* severe medical comorbidity impairing daily activities (inability to go climb three floors without assistance and stopping)
* Body Mass Index over 40
* unacceptably high risk of surgery due to severe medical comorbidities
* severe substance abuse
* patient is retired
* age is less than 18 or more than 65
* patient required a fasciotomy due to acute compartment syndrome during or after index surgery
* inability to walk before fracture or a daily need of walking aid, such as crutches

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Return to work | 3 months
  Rate of return to work
Physical component summary | 3 months
  Physical component summary of the SF-36 questionnaire

SECONDARY OUTCOMES:
Return to work | 6 months
  Rate of return to work
Return to work | 12 months
  Rate of return to work
Physical component summary | 6 months
  Physical component summary of the SF-36 questionnaire
Physical component summary | 12 months
  Physical component summary of the SF-36 questionnaire
Total sick leave | 12 months
  Overall length of sick leave
Lower extremity functional scale | 3 months
  Measurement of lower extremity function with a scale from 0 (worst) to 100 (best).
Lower extremity functional scale | 6 months
  Measurement of lower extremity function with a scale from 0 (worst) to 100 (best).
Lower extremity functional scale | 12 months
  Measurement of lower extremity function with a scale from 0 (worst) to 100 (best).
Lower extremity functional scale | 24 months
  Measurement of lower extremity function with a scale from 0 (worst) to 100 (best).
36-Item Short Form Survey | 3 months
36-Item Short Form Survey | 6 months
36-Item Short Form Survey | 12 months
36-Item Short Form Survey | 24 months
Tegner activity level scale | 3 months
  Method of grading work and sporting activities
Tegner activity level scale | 6 months
  Method of grading work and sporting activities
Tegner activity level scale | 12 months
  Method of grading work and sporting activities
Tegner activity level scale | 24 months
University of California and Los Angeles activity level scale | 3 months
  Method of grading work and sporting activities
University of California and Los Angeles activity level scale | 6 months
  Method of grading work and sporting activities
University of California and Los Angeles activity level scale | 12 months
  Method of grading work and sporting activities
University of California and Los Angeles activity level scale | 24 months
  Method of grading work and sporting activities
Complications | 6 weeks
  Surgery related complications
Complications | 3 months
  Surgery related complications
Complications | 6 months
  Surgery related complications
Complications | 12 months
  Surgery related complications
Complications | 24 months
  Surgery related complications

OTHER OUTCOMES:
Total ground force during gait | 3 weeks
  Measurement of lower leg activity using pressure insoles

CONTACTS AND LOCATIONS:
Overall Officials: Aleksi Reito, Assoc prof, Principal Investigator — Tampere University Hospital
Locations (3):
- Finland (3):
  - Central Finland Hospital Nova, Jyväskylä, Central Finland
  - Tampere Univeristy Hospital, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland

IPD SHARING:
Plan to Share IPD: Yes
IDP can be shared based on a reasonable request
Access Criteria: On a reasonable request along with a research plan.